CLINICAL TRIAL: NCT01930006
Title: Phase 1 Single Dose 2-Way Crossover Comparative Bioavailability Study Of Two Oral Formulations Of MGCD265 In Healthy Male And Female Subjects - Fasting State
Brief Title: Safety Study of Two Oral Formulations of MGCD265 Administered in Healthy Subjects in the Fasting State
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mirati Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 265-106
Record Dates: First submitted 2013-08-23; First posted 2013-08-28 (Estimated); Last update posted 2015-01-08 (Estimated); Status verified 2015-01

CONDITIONS: Advanced Malignancies
Keywords: c-Met; VEGFR; Ron; Cancer; Tumor; Safety; Phase 1
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MGCD265 (Experimental)
  Interventions: Drug: MGCD265

INTERVENTIONS:
Drug: MGCD265

SUMMARY:
In this study two MGCD265 oral formulations at dose level of 100 mg are administered to healthy male and female subjects under fasting conditions.

DETAILED DESCRIPTION:
The objective of this study is to compare the rate and extent of absorption of two MGCD265 oral formulations at a dose level of 100 mg administered to healthy male and female subjects under fasting conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female subjects ≥18 to ≤55 years of age who are willing and able to provide informed consent prior to performing any study related procedures
2. Females of childbearing potential who are using a stable contraceptive method at least 30 days prior to screening and who are willing to use one of the following acceptable birth control methods until 30 days after the last dose of study drug:

   1. Abstinence
   2. Hormonal contraceptives (birth control pills, injectable/ implantable/ insertable hormonal birth control products, transdermal patch) for at least 3 months prior to the first dose of the study drug and male condom and intravaginal spermicide
   3. Intra-uterine contraceptive device (IUD) in place for at least 3 months prior to the first dose of study drug plus spermicide and male condom
   4. Male condom and diaphragm plus spermicide;
   5. Male condom and cervical cap plus spermicide;
   6. Surgical sterilization of the partner(s) (vasectomy for 6 months minimum prior to the first dose of study drug)
3. Female subjects will be considered of non childbearing potential and eligible if one of the following condition is met:

   1. Amenorrhea for at least 1 year, with confirmation by a follicle-stimulating hormone (FSH ≥ 40 mIU/mL)
   2. Hysterectomy
   3. Bilateral oophorectomy
   4. Bilateral tubal ligation
4. Male subjects must agree to be abstinent or use the following acceptable contraception methods in collaboration with their female partner from the time of taking the first dose until 3 months after the last dose of study drug:

   1. Male condom and intravaginal spermicide plus hormonal contraceptives (birth control pills, injectable/ implantable/ insertable hormonal birth control products, transdermal patch) in use for at least 3 months
   2. Male condom and IUD in place for at least 3 months plus spermicide;
   3. Male condom and diaphragm plus spermicide
   4. Male condom and cervical cap plus spermicide
   5. Vasectomy for 6 months minimum prior to the first dose of study drug

   Male subjects also agree to not donate sperm from the time of taking the first dose of study drug until 3 months after the last dose of study drug
5. Subject with a body mass index (BMI) of 18.0 to 32.0 kg/m2 at screening
6. Subject is a current non-smoker and has not used any nicotine containing product within 3 months prior to screening
7. Subjects who are considered generally healthy upon completion of medical history, physical examination, vital signs, screening laboratory results and screening ECG as judged by the investigator
8. Subjects who are willing and able to comply with the visit schedule, treatment plan, laboratory tests, pharmacokinetic sampling schedule and other study procedures

Exclusion Criteria:

1. Females who are pregnant or are breast feeding
2. History of significant hypersensitivity reaction to any substance or drug
3. Clinically relevant history or evidence of significant gastrointestinal, hepatic, renal, endocrine, pulmonary, neurological, psychiatric, cardiovascular, hematologic, dermatologic, immunologic disease or any other condition known to interfere with the absorption, distribution, metabolism or distribution of drugs that in the opinion of the investigator would jeopardize the safety of the subject or impact validity of study results
4. Clinically significant vital signs in the opinion of the investigator at screening or prior to study drug administration
5. History of clinically significant cardiovascular illness including but not confined to: angina pectoris or myocardial infarction, coronary or peripheral artery bypass graft, congestive heart failure, or clinically significant cardiac arrhythmia in the opinion of the investigator
6. History of clinically significant thrombotic or hemorrhagic events (including but not confined to stroke and transient ischemic attacks); history of bleeding diathesis or coagulopathy; history or presence of gastrointestinal or other conditions with risk of perforation; presence of a non-healing wound, ulcer or fracture in the opinion of the investigator
7. Presence of out-of-range cardiac interval (PR < 110 msec, PR > 200 msec, QRS < 60 msec, QRS >110 msec and QTcF > 450 msec) at screening or the pre-dose ECG or other clinically significant ECG abnormalities in the opinion of the investigator
8. History of regular alcohol consumption exceed 7 drinks for females and 14 drinks per week for males within 6 months of screening or a positive alcohol breath test at screening and prior to study drug administration
9. History of significant drug abuse within one year prior to screening
10. Any clinically significant illness or surgery in the previous 30 days before day 1 of this study
11. Use of any enzyme-modifying drugs, including strong inhibitors of cytochrome P450 (CYP) enzymes (such as cimetidine, fluoxetine, quinidine, erythromycin, ciprofloxacin, fluconazole, ketoconazole, diltiazem and HIV antivirals) and strong inducers of CYP enzymes (such as barbiturates, carbamazepine, glucocorticoids, phenytoin, rifampin and St John's Wort), in the previous 30 days before day 1 of this study
12. Use of any drugs known to induce or inhibit hepatic metabolism (inducers such as rifampin, barbiturates, carbamazepine, phenytoin, glucocorticoid, omeprazole; inhibitors such as antidepressants (SSRI), cimetidine, diltiazem, macrolides, imidazoles, neuroleptics, verapamil, fluroquinolones, antihistamines) in the previous 30 days before day 1 of the study
13. Use of any other prescription medications in the previous 14 days before day 1 of this study
14. Use of any over-the-counter (OTC) products including cold preparations, multivitamins and dietary supplements used for therapeutic benefits and antacid preparations in the previous 7 days before day 1 of this study
15. Use of Acetylsalicylic Acid (ASA) or NSAIDs (or any product containing ASA or NSAIDs) in the previous 7 days before day 1 of this study
16. Use of MAO inhibitors within 30 days of day 1 of the study
17. Positive urine drug screen or urine cotinine test at screening and prior to study drug administration
18. Positive results to HIV, HBsAg or anti-HCV tests at screening
19. Subjects who took an Investigational Product (in another clinical trial) in the previous 30 days (90 days for biologics) before day 1 of this study
20. Donation of plasma within 7 days prior to dosing. Any donation/loss of blood or blood products within 3 months of the screening visit
21. Prior exposure to MGCD265

No subjects will be allowed to enroll in this study more than once (i.e. if the study is conducted with more than 1 group).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2013-08; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
To assess the bioavailability of two MGCD265 formulations. | Two months
  To compare the rate and extent of absorption of two MGCD265 oral formulations at dose level of 100 mg administered as 1 x 100 mg oral dose (Formulation A) and 2 x 50 mg oral dose (Formulation B) under fasting conditions.

CONTACTS AND LOCATIONS:
Locations (1):
- Vince & Associates Clinical Research, Inc., Overland Park, Kansas, United States